CLINICAL TRIAL: NCT05722054
Title: Trained and Heterologous Induced-immune Responses to Tropical Infectious Diseases: Selection and Validation of Immune Assays in Children Aged 1-12 Years Living in Lambaréné, Gabon
Brief Title: Trained and Heterologous Induced-immune Responses to Tropical Infectious Diseases
Acronym: TSH-IMMO
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Centre de Recherche Médicale de Lambaréné (Other)
Responsible Party: Sponsor
Other Study IDs: CEI-007/2022
Record Dates: First submitted 2022-12-03; First posted 2023-02-10 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Tropical Infectious Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, Plasma, Whole blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Incidence of tropical infectious diseases: All study participants will be followed up for 12 months through active and passive detection visits. Active detection takes place every month for all pathogens except for P. falciparum which is detected every two weeks.
  Interventions: Other: Diagnostic tests
- Healthy and equilibrate diet: One-fourth of the study participants will be randomly assigned to receive an equilibrate diet for 21 days comprising breakfast, lunch and educational recommendations for an equilibrate diet
  Interventions: Other: Equilibrate diet
- In vitro: 30 to 50 participants selected from the study population. The in vitro study procedures are performed at the screening visit and every two months+/- 1, and when an active case of tropical infection occurs
  Interventions: Other: Diagnostic tests
- Adaptive in vitro: 100 to 150 selected participants. The adaptive in vitro study procedures are performed at the screening visit and every two months+/- 1 and when an active case of tropical infection occurs.
  Interventions: Other: Diagnostic tests
- Ex vivo: All study participants. The ex vivo are performed at the screening visit and every two months+/- 1 and when an active case of tropical infection occurs.
  Interventions: Other: Diagnostic tests

INTERVENTIONS:
Other: Diagnostic tests — Blood smears; rapid diagnostic tests; complete blood counts with differential; "leucoconcentration"; urine examination; nasal/throat swabs, stool examination.
  Groups: Adaptive in vitro; Ex vivo; In vitro; Incidence of tropical infectious diseases
Other: Equilibrate diet — Nutritionally-balanced Alimentation
  Groups: Healthy and equilibrate diet

SUMMARY:
Validation of ex vivo immune assays that are surrogates of complex in vitro assays and animal models studies to identify the occurrence, strength, and kinetics of trained and heterologous immunity may significantly impact public health. In this study, the investigators translate findings from systems biology approaches into contextualized in vitro and ex vivo assays in children living in settings where tropical infectious diseases are highly prevalent. The investigators first reproduce the Vitro assays using culture of monocytes, co-culture of T cells and dendritic cells. Based on data from contextualized assays, the investigators will select, test, and validate candidates' surrogate markers of trained immunity and heterologous immunity.

The TSH-IMMO is a prospective cohort study. Participants aged 1 to 12 years and living in Lambaréné, Gabon, will be recruited.

DETAILED DESCRIPTION:
Overview of the study The investigators will conduct a prospective cohort study. Participants aged 1 to 12 years will be recruited and undergo baseline clinical and biological assessments and receive a curative dose of either artemether-Lumefantrine or dihydroartemisinin-piperaquine to clear any existing P.falciparum parasitemia. Clearance of parasites will be confirmed 3 weeks later by PCR, and only participants with negative PCR will be definitively enrolled for the longitudinal follow up. Both active and passive case detection will ensure that a high proportion of infections in the cohort is captured. In addition, participants with any other active tropical infections except the viral infections will be treated within the three weeks according to national treatment guidelines.

For the active follow up, participants will be actively seen every month for supervised clinical evaluations and to collect blood samples for detecting tropical infections according to the gold-standard test, PCR and serodiagnosis. Participants will be followed passively in parallel to monthly visits; diagnosis of tropical infectious diseases will be performed upon clinical evaluation. Participants will be followed for 12 months.

Screening The screening visit aims to determine subject eligibility for study participation. Screening procedures follow Informed consent procedures, clinical assessments, diagnosis of tropical infections, and hemoglobin level. Baseline immune responses will also be performed.

P. falciparum parasite clearance and treatment of other tropical infections. All children, irrespective of malaria parasite status, will receive a curative antimalarial dose to clear any existing parasitaemia. Children will be treated according to local guidelines when found with an active infection of M. perstans, Loa, loa, Dengue virus, Chikungunya virus, SARS-CoV2, resistant bacteria, S. haematobium, N. americanus, Ascaris lumbricoides, Trichuris trichiura, S. stercoralis, protozoa spp.

Follow up of enrolled participants The study will combine active and passive case detection surveys with meeting study objectives and capturing full episodes of tropical infections from enrolled study participants. In addition, studies on trained and heterologous immunity will take place.

For P. falciparum

The following procedures will be followed:

* Questioning for symptoms of malaria, prevention measures, fever and medication since the previous visit
* Temperature measurement
* Perform careful clinical examination and syndrome summary
* Venous blood sample collection
* Blood smear
* Rapid diagnostic test (RDT)
* Parasite DNA extraction

Children with fever or history of fever will be referred to the local health centre:

* Rapid diagnostic test (RDT) in case of history of fever in 24 H/ fever (Axillary temperature ≥37.5°C/Tympanic ≥38°C or Forehead temperature ≥37.5°C using non- contact infrared thermometer) (50 μL)
* Confirmed malaria cases will follow these procedures:

  o Treatment as per government guidelines.
* Others causes of fever will be managed according to the national guidelines.

For other pathogens The detection takes place every month at the clinic of CERMEL.

* Questioned for symptoms of disease induced by the targeted pathogens, prevention measures, fever and medication since the previous visit
* Perform careful clinical examination and syndrome summary
* EDTA for RDT, blood smear, complete blood count, microfilaria (microscopy and Leucoconcentration), DNA and RNA extraction
* Urine sample for S. haematobium, bacteria
* Nasal and throat swabs for SARS-CoV2
* Throat swabs for bacteria
* Stool examination for helminths and protozoa

For trained and heterologous immunity Human DNA extraction; cell cultures and analyses; seroprevalence studies

ELIGIBILITY:
Inclusion Criteria:

* Healthy children aged 1 to 12 years
* Residence in the study area or surroundings for the period of the study
* Written informed consent from parents/legally acceptable representatives and an assent for children (age will depend on local country regulations)

Exclusion Criteria:

* Complicated symptomatic malaria (defined according to standard World Health Organization criteria)
* Anaemia (Hb<7g/dL),
* Any (chronic) illness that requires immediate clinical care
* Family history of sudden death or of congenital or clinical conditions known to prolong QTcB or QTcF interval or e.g. family history of symptomatic cardiac arrhythmias, with clinically relevant bradycardia or severe cardiac disease
* Any treatment which can induce a lengthening of Q.T. interval
* Known history of hypersensitivity or allergic reactions to piperaquine or other aminoquinolines and Lumefantrine
* Receipt of any blood transfusion or immunoglobulins within 3 months
* Known history of hypersensitivity or allergic reactions to artesunate
* Severe malnutrition (weight-for-height being below -3 standard deviation or less than 70% of median of the NCHS/WHO normalized reference values).
* Weight below 5 kg
* Current participation in malaria vaccine trials
* Current active participation in any trial involving administration of investigational drug.
* Any severe drug-drug interactions, antimalarial, antihelminth and antibiotics

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The TSH-IMMO study will be conducted at the Centre de Recherches Médicales de Lambaréné (CERMEL), Gabon. CERMEL has established a demographic and health surveillance system that covers Lambaréné and a radius of about 70 Km away in both North and South directions.
  About 8,000 households are in the surveillance system. Our surveillance system has estimated that 30,000 inhabitants live in the area and about 27% are aged 1-12 years old. There are 1 to 24 inhabitants in the households, with a median of 3-4 inhabitants per household.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Incidence, morbidity, and transmission of tropical infectious diseases | At 12 months
  To assess the incidence/ transmission of P. falciparum, M. perstans, Loa, loa, Dengue virus, Chikungunya virus, SARS-CoV2, resistant bacteria, S. haematobium, N. americanus, Ascaris lumbricoides, Trichuris trichiura, S. stercoralis, protozoa spp

IPD SHARING:
Plan to Share IPD: Undecided